CLINICAL TRIAL: NCT07225556
Title: A Phase 1, Randomized, Placebo-Controlled, Single Ascending Dose-Escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY4167586 in Participants With Obesity or Overweight Who Are Otherwise Healthy
Brief Title: A Study of LY4167586 in Participants With Obesity or Overweight Who Are Otherwise Healthy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 27659; J6L-MC-YIAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-10-20; First posted 2025-11-06 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY4167586 (Cohorts A1 to A6) (Experimental): LY4167586 administered subcutaneously (SC)
  Interventions: Drug: LY4167586
- LY4167586 (Cohorts A1 to A6) Placebo (Placebo Comparator): LY4167586 administered SC
  Interventions: Drug: Placebo
- LY4167586 (Cohort B) (Experimental): LY4167586 administered intravenously (IV)
  Interventions: Drug: LY4167586

INTERVENTIONS:
Drug: LY4167586 — Administered SC
  Arms: LY4167586 (Cohorts A1 to A6)
Drug: Placebo — Administered SC
  Arms: LY4167586 (Cohorts A1 to A6) Placebo
Drug: LY4167586 — Administered IV
  Arms: LY4167586 (Cohort B)

SUMMARY:
The purpose of this study is to look at how safe and well-tolerated LY4167586 is in participants with obesity or overweight who are otherwise healthy. Blood tests will be performed to check how much LY4167586 gets into the bloodstream and how long it takes the body to eliminate it following a single administration. Participation in the study will last approximately 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 21 for Singapore site
* Have a body mass index (BMI) between 27.0 kilogram per square meter (kg/m²) and 35.0 kg/m², inclusive
* Have had a self-reported stable weight for 3 months prior to screening (less than approximately 5 percent [%] body weight change)

Exclusion Criteria:

* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal (GI), endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs, or of constituting a risk when taking the study drug, or of interfering with the interpretation of data.
* Is an individual of childbearing potential (IOCBP)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number and Incidence of Serious Adverse Events (SAEs) | Baseline to study completion (up to 29 weeks)
  A summary of SAEs regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) | Predose on Day 1 through end of the Follow-up Period (Week 25)
  PK: Cmax of LY4167586
PK: Time of Maximum Drug Concentration (tmax) | Predose on Day 1 through end of the Follow-up Period (Week 25)
  PK: tmax of LY4167586
PK: Area Under the Concentration Versus Time Curve (AUC) | Predose on Day 1 through end of the Follow-up Period (Week 25)
  PK: AUC of LY4167586

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Fortrea Clinical Research Unit, Madison, Wisconsin, United States
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No